CLINICAL TRIAL: NCT03046524
Title: Parathyroid Cancer Versus Atypical Parathyroid Neoplasm; Investigating Their Clinical Characteristics and Biological Behavior
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA15-0808
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Parathyroid Carcinoma; Parathyroid Neoplasm
Keywords: Parathyroid Carcinoma; Parathyroid Neoplasm; Chart Review
MeSH Terms: conditions — Parathyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parathyroid Carcinoma: Charts from participants with histopathological diagnosis of parathyroid carcinoma.
  Interventions: Other: Chart Review
- Atypical Parathyroid Neoplasm: Charts from participants with parathyroid tumors with some atypical features found in parathyroid carcinoma, but not enough histologic criteria to make the diagnosis of parathyroid carcinoma.
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — Data between the years of 1/1/2002 and 12/31/2013 analyzed.

SUMMARY:
Objectives:

1. Identify the clinical characteristics of parathyroid (PTH) cancer and PTH atypical neoplasms
2. Investigate if PTH carcinoma and atypical neoplasm present a biological behaviour and have a different impact on the health of the patients

DETAILED DESCRIPTION:
Data between the years of 1/1/2002 and 12/31/2013 will be analyzed. The medical records of all adult patients that had a parathyroidectomy for primary PHPT in MD Anderson Cancer Center will be screened in order to identify patients that had a histopathological diagnosis of parathyroid carcinoma or atypical parathyroid neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* All patients from MDACC diagnosed with PHPT that have a histopathological diagnosis of PTH carcinoma or atypical parathyroid neoplasm between the years 1/1/2002 and 12/31/2013

Exclusion Criteria:

* Pediatric patients
* Cases with incomplete records
* Patients where the follow-up will be less than six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical records of all adult patients that had a parathyroidectomy for primary PHPT in MD Anderson Cancer Center between the years of 1/1/2002 and 12/31/2013.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Information Collected on Clinical Characteristics of Parathyroid (PTH) Cancer and PTH Atypical Neoplasms by Conducting a Retrospective Chart Review | 5 years
Information Collected on PTH Carcinoma's Biological Behaviour and Impact on the Health of the Patients by Conducting a Retrospective Chart Review | 5 years
Information Collected on Atypical Neoplasm's Biological Behaviour and Impact on the Health of the Patients \by Conducting a Retrospective Chart Review | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org